CLINICAL TRIAL: NCT00213434
Title: Prospective Evaluation of Mandibular Advancement by Herbst Device in the Treatment of Moderate Obstructive Sleep Apnea Syndrome
Brief Title: Evaluation of a Mandibular Advancement Device in the Treatment of Obstructive Sleep Apnea Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2000/055/HP
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2013-06-26 (Estimated); Status verified 2013-06

CONDITIONS: Obstructive Sleep Apnea
Keywords: prospective; randomized; polysomnography; orthodontic appliance, removable
MeSH Terms: conditions — Sleep Apnea, Obstructive

INTERVENTIONS:
Device: Herbst oral appliance

SUMMARY:
The purpose of this study is to determine if the mandibular advancement by Herbst device is effective in the treatment of moderate obstructive sleep apnea patients.

ELIGIBILITY:
Inclusion Criteria:

* Moderate sleep apnea syndrome (10 < Respiratory Disorder Index < 30)
* Body mass index (BMI) < 35 Kg/m2
* Able to give their informed consent

Exclusion Criteria:

* Pregnant women
* Professional drivers requiring continuous positive airway pressure (CPAP) treatment
* Psychiatric disorders, and patients unable to realise to study
* Severe respiratory pathology which could interfere with the study
* Morpheic epilepsy
* Benzodiazepines intake
* Chronic nasal obstruction
* Ear, nose, and throat (ENT) pathology requiring surgery
* Previous uvulopalatoplasty surgery
* Temporomandibular joint pathology
* Gum disease
* Insufficient number of teeth to apply the oral appliance
* Mobile teeth

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-11; Primary Completion 2004-12 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Comparison of polysomnographic data after 3 months of treatment by oral appliance in 2 groups: one with Herbst device adjusted in maximal mandibular advancement and a placebo group

SECONDARY OUTCOMES:
Efficacy on clinical symptoms
Tolerance of the oral appliance
Identification of predictive factors of efficacy
Feasibility of this therapeutic method

CONTACTS AND LOCATIONS:
Overall Officials: PORTIER PF Florence, MD, Principal Investigator — University Hospital, Rouen
Locations (1):
- CHU de ROUEN, Rouen, France